CLINICAL TRIAL: NCT07145918
Title: An Adaptive Two-part Randomized, Double Blind, Placebo-controlled Phase 2 Study to Assess the Safety, Tolerability, Pharmacokinetics, and Efficacy of Emraclidine in Participants With Schizophrenia
Brief Title: A Study to Assess Adverse Events, Change in Disease Activity, and How Oral Emraclidine Moves Through the Body in Adult Participants With Schizophrenia
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: M25-522
Record Dates: First submitted 2025-08-22; First posted 2025-08-28 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Schizophrenia
Keywords: Schizophrenia; ABBV-1231
MeSH Terms: conditions — Schizophrenia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (4):
- Emraclidine Part A (Experimental): Participants will be assigned to received one of multiple ascending doses of oral emraclidine for 14 or up to 21 days, followed by a 30-day safety follow-up period.
  Interventions: Drug: Emraclidine
- Placebo-Part A (Experimental): Participants will be assigned to received one of multiple ascending doses of oral placebo for 14 or up to 21 days, followed by a 30-day safety follow-up period.
  Interventions: Drug: Placebo
- Emraclidine-Part B (Experimental): Participants will receive oral emraclidine for 42 days followed by a 30-day safety follow-up period.
  Interventions: Drug: Emraclidine
- Placebo-Part B (Experimental): Participants will receive placebo for 42 days followed by a 30-day safety follow-up period.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Emraclidine — Oral Tablets
  Arms: Emraclidine Part A; Emraclidine-Part B
Drug: Placebo — Oral Tablets
  Arms: Placebo-Part A; Placebo-Part B

SUMMARY:
Schizophrenia is a common and severe psychiatric illness characterized by extreme disturbances of cognition and thought, affecting language, perception and sense of self. This study will assess adverse events, change in disease activity, and how oral emraclidine moves through the body in adult participants with schizophrenia

Emraclidine is an investigational drug being developed for the treatment of schizophrenia. Participants are placed in one of two parts, Part A or Part B, where each group will receive a different treatment. Participants will receive either oral emraclidine or placebo. Approximately 268 participants will be enrolled across roughly 32 sites in the United States.

Participants in Part A will be assigned to one of multiple ascending doses of emraclidine or placebo administered orally for 14 days or up to 21 days. Participants in Part B will receive Emraclidine or placebo administered orally for up to 42 days. Participants will be followed for 30 days after the last dose of the study drug.

There may be higher treatment burden for participants in this trial compared to their standard of care. Participants will attend regular visits during the study at a hospital or clinic. The effect of the treatment will be checked by medical assessments, blood tests, checking for side effects and completing questionnaires.

ELIGIBILITY:
Inclusion Criteria:

* BMI within 18 to 40 kg/m2 (inclusive of both values), and body weight > 50 kg (110 lbs).
* (Part A only): Positive and Negative Syndrome Scale (PANSS) total score < 80 at Screening and at Baseline
* (Part B only): Participant experiencing an acute exacerbation of psychotic symptoms with onset less than 2 months prior to Screening
* (Part B only): Participant must have a PANSS total score from 80 to 120, inclusive, at Screening and at Baseline
* (Part B only): Participant MUST have a score of ≥ 4 (moderate or greater) for ≥ 2 of the following PANSS Positive Scale items at Screening and at Baseline
* (Part B only): Participant must have a Clinical Global Impression of Severity (CGIS) score ≥ 4 (at least moderately ill) at Screening and Baseline

Exclusion Criteria:

* Any primary DSM-5 disorder other than schizophrenia (current nicotine use disorder and caffeine use disorder are allowed) within 12 months before Screening.
* History of clozapine exposure.
* History of treatment resistance to schizophrenia medications, defined as failure to respond to 2 or more adequate courses of pharmacotherapy (a minimum of 4 weeks at an adequate dose per the label) within the last 12 months

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 268 (Estimated)
Dates: Start 2025-08-04 (Actual); Primary Completion 2028-02 (Estimated); Study Completion 2028-02 (Estimated)

PRIMARY OUTCOMES:
Number of Participants with Adverse Events (AEs) | Up to approximately 74 days
  An adverse event (AE) is defined as any untoward medical occurrence in a patient or clinical investigation participant administered a pharmaceutical product which does not necessarily have a causal relationship with this treatment. The investigator assesses the relationship of each event to the use of study.
Part A Only-Maximum Observed Plasma Concentration (Cmax) of Emraclidine | Up to approximately 24 days
  Cmax of Emraclidine
Part A Only-Time to Cmax (Tmax) of Emraclidine | Up to approximately 24 days
  Tmax of Emraclidine
Part A Only-Area Under the Concentration-Time Curve from Time 0 to Time t (AUCt) of Emraclidine | Up to approximately 24 days
  AUCt of Emraclidine
Part A Only-Area under the plasma concentration-time curve over the dosing interval (AUCtau) of Emraclidine | Up to approximately 24 days
  AUCtau of Emraclidine
Part A Only-Maximum metabolite concentration (MRCmax) of Emraclidine | Up to approximately 21 days
  MRCmax of Emraclidine
Part A Only- Area under the metabolite concentration-time curve over the dosing interval (MRAUCtau) of Emraclidine | Up to approximately 21 days
  MRAUCtau of Emraclidine
Part A Only- Minimum plasma concentration (Cmin) of Emraclidine | Up to approximately 21 days
  Cmin of Emraclidine
Part A Only-Average plasma concentration (Cavg) of Emraclidine | Up to approximately 21 days
  Cavg of Emraclidine
Part A Only- Terminal Phase Elimination Half-Life (t1/2) of Emraclidine | Up to approximately 21 days
  Terminal phase elimination half-life of Emraclidine
Part A Only-Terminal elimination rate constant (λz) of Emraclidine | Up to approximately 21 days
  λz of Emraclidine
Part A Only-Apparent Clearance of Drug from Plasma (CL/F) of Emraclidine | Up to approximately 21 days
  CL/F of Emraclidine
Part A Only-Apparent Volume of Distribution DuringTerminal Phase (Vz/F) of Emraclidine | Up to approximately 21 days
  Vz/F of Emraclidine
Part A Only-Peak-to-trough ratio (PTR) of Emraclidine | Up to approximately 21 days
  PTR of Emraclidine
Part A Only- Accumulation ratio for Cmax (RacCmax) of Emraclidine | Up to approximately 21 days
  RacCmax of Emraclidine
Part A Only-Accumulation ratio for AUCta (RacAUCtau) of Emraclidine | Up to approximately 21 days
  RacAUCta of Emraclidine
Part A Only-Maximum Observed Plasma Concentration (Cmax) of Metabolite (CV-0000364) | Up to approximately 24 days
  Cmax of Metabolite (CV-0000364)
Part A Only-Time to Cmax (Tmax) of Metabolite (CV-0000364) | Up to approximately 24 days
  Tmax of Metabolite (CV-000036)
Part A Only-Area under the plasma concentration-time curve over the dosing interval (AUCtau) of Metabolite (CV-000036) | Up to approximately 24 days
  AUCtau of Metabolite (CV-000036)
Part A Only-Area Under the Concentration-Time Curve from Time 0 to Time t (AUCt) Metabolite (CV-000036) | Up to approximately 24 days
  AUCt of Metabolite (CV-000036)
Part A Only-Maximum metabolite concentration (MRCmax) of Metabolite (CV-000036) | Up to approximately 21 days
  MRCmax of Metabolite (CV-000036)
Part A Only- Area under the metabolite concentration-time curve over the dosing interval (MRAUCtau) of Metabolite (CV-000036) | Up to approximately 21 days
  MRAUCtau of Metabolite (CV-000036)
Part B Only-Change from Baseline in Positive and Negative Syndrome Scale (PANSS) total score | Up to approximately week 6
  PANSS is a 30-item clinician-reported rating scale which assesses both the positive and negative symptom syndromes of patients with schizophrenia. The PANSS consists of 3 subscales containing a total of 30 symptom constructs. For each symptom construct, severity is rated on a 7-point scale, with a score of 1 indicating the absence of symptoms and a score of 7 indicating extremely severe symptoms.

SECONDARY OUTCOMES:
Part B Only-Change from Baseline in in Clinical Global Impression of Severity (CGIS) score | Up to approximately Week 6
  CGIS is a single, clinician-reported item that measures the clinician's impression of a participant's current anxiety severity considering their total clinical experience with the patient population. The measure uses a 7-point Likert rating scale with responses ranging from "normal, to at all ill" (1) to "among the most extremely ill patients" (5), with higher scores indicating greater anxiety severity.
Part B Only-Change from Baseline in Positive and Negative Syndrome Scale (PANSS) total score | Up to approximately 74 days
  PANSS is a 30-item clinician-reported rating scale which assesses both the positive and negative symptom syndromes of patients with schizophrenia. The PANSS consists of 3 subscales containing a total of 30 symptom constructs. For each symptom construct, severity is rated on a 7-point scale, with a score of 1 indicating the absence of symptoms and a score of 7 indicating extremely severe symptoms.
Part B Only-Change from Baseline in in Clinical Global Impression of Severity (CGIS) score | Up to approximately 53 days
  CGIS is a single, clinician-reported item that measures the clinician's impression of a participant's current anxiety severity considering their total clinical experience with the patient population. The measure uses a 7-point Likert rating scale with responses ranging from "normal, to at all ill" (1) to "among the most extremely ill patients" (5), with higher scores indicating greater anxiety severity.
Part B Only-Number of Participants achieving ≥ 30% improvement in PANSS total score | Up to approximately week 6
  PANSS is a 30-item clinician-reported rating scale which assesses both the positive and negative symptom syndromes of patients with schizophrenia. The PANSS consists of 3 subscales containing a total of 30 symptom constructs. For each symptom construct, severity is rated on a 7-point scale, with a score of 1 indicating the absence of symptoms and a score of 7 indicating extremely severe symptoms.
Part B Only-Number of Participants achieving remission (PANSS total score ≤ 60) | Up to approximately week 6
  PANSS is a 30-item clinician-reported rating scale which assesses both the positive and negative symptom syndromes of patients with schizophrenia. The PANSS consists of 3 subscales containing a total of 30 symptom constructs. For each symptom construct, severity is rated on a 7-point scale, with a score of 1 indicating the absence of symptoms and a score of 7 indicating extremely severe symptoms.

CONTACTS AND LOCATIONS:
Overall Officials: ABBVIE INC., Study Director — AbbVie
Locations (7):
- United States (7):
  - Woodland International Research Group /ID# 275747, Little Rock, Arkansas
  - Collaborative Neuroscience Research - Garden Grove /ID# 273005, Garden Grove, California
  - California Clinical Trials Medical Group - Parexel /ID# 275751, Glendale, California
  - Cbh Health - Gaithersburg /ID# 272932, Gaithersburg, Maryland
  - Cenexel Hassman Research Institute (Hri) /ID# 276128, Marlton, New Jersey
  - Community Clinical Research - Austin - Cross Park Drive /ID# 272977, Austin, Texas
  - Pillar Clinical Research - Richardson /ID# 275715, Richardson, Texas

IPD SHARING:
Plan to Share IPD: Yes
AbbVie is committed to responsible clinical trial data sharing. This includes access to anonymized, individual and trial-level data (analysis data sets), as well as other information.
Supporting Information: Study Protocol, SAP
Time Frame: For details on when studies are available for sharing, visit https://vivli.org/ourmember/abbvie/
Access Criteria: To learn more about the process, or to submit a request, visit the following link https://www.abbvieclinicaltrials.com/hcp/data-sharing/
URL: https://vivli.org/ourmember/abbvie/

REFERENCES:
- See also: Related Info — https://www.abbvieclinicaltrials.com/study/?id=M25-522